CLINICAL TRIAL: NCT01830881
Title: An Evaluation of Oral Midazolam for Anxiety and Pain in First-trimester Surgical Abortion: a Randomized Controlled Trial
Brief Title: Evaluation of Oral Midazolam in First-trimester Surgical Abortions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lisa Bayer, MD MPH, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 9064
Record Dates: First submitted 2013-04-03; First posted 2013-04-12 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Pain; Anxiety; Nausea
Keywords: pain; anxiety; surgical abortion; midazolam; benzodiazepine
MeSH Terms: conditions — Pain; Anxiety Disorders; Nausea | interventions — Midazolam; Ibuprofen; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo-cherry syrup and ibuprofen (Placebo Comparator): 5 mL oral placebo-cherry syrup and 800 mg oral ibuprofen 30-60 minutes prior to procedure 20 mL injection 1% lidocaine without epinephrine
  Interventions: Drug: Ibuprofen; Other: Placebo-Cherry syrup; Drug: Lidocaine
- Midazolam and ibuprofen (Active Comparator): 5 mL oral midazolam oral syrup (2 mg/mL) and 800 mg oral ibuprofen 30-60 minutes prior to procedure 20 mL injection 1% lidocaine without epinephrine
  Interventions: Drug: Midazolam; Drug: Ibuprofen; Drug: Lidocaine

INTERVENTIONS:
Drug: Midazolam — 5 mL oral midazolam oral syrup (2 mg/mL) 30-60 minutes prior to procedure
  Other Names: Versed
  Arms: Midazolam and ibuprofen
Drug: Ibuprofen — 800 mg oral ibuprofen 30-60 minutes prior to procedure
  Other Names: Motrin
Other: Placebo-Cherry syrup — 5 mL oral placebo-cherry syrup 30-60 minutes prior to procedure
  Other Names: placebo cherry syrup
  Arms: placebo-cherry syrup and ibuprofen
Drug: Lidocaine — injection of 20 mL 1% lidocaine without epinephrine
  Other Names: lidocaine injection

SUMMARY:
The purpose of this study is to determine the level of pain, anxiety and side effects that women experience with a surgical abortion and the effect that the anti-anxiety medication, midazolam, might have when used along with ibuprofen and a paracervical block (PCB) instead of the standard pain treatment of only ibuprofen and a PCB.

DETAILED DESCRIPTION:
Women in the study will be randomized to receive either midazolam or placebo. Every participant will still receive the standard oral medications for pain (ibuprofen) as well as an injection of numbing medicine (lidocaine) near the cervix (PCB). The co-primary outcomes are patient perception of anxiety and pain with uterine aspiration reported on a 100 mm visual analogue scale (VAS). Secondary outcomes include reported anxiety and pain at time points before, during, and after the procedure, as well as subject satisfaction with anxiety and pain control and overall abortion experience. Due to the dose-dependent anterograde amnesic effect of midazolam, we will also investigate the effects on memory and recall, which has not previously been studied. In addition, we will also collect data on side effects frequently associated with oral midazolam such as nausea and sleepiness. Women will also be responsible for completing a one-page survey 1-3 days after the procedure visit and return it by mail using a pre-addressed and stamped envelope.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Voluntarily requesting surgical pregnancy termination
* Pregnancy with intrauterine gestational sac between 6 0/7 and 10 6/7 weeks gestation, dated by ultrasound
* Eligible for suction aspiration
* English or Spanish speaking
* Good general health
* Able and willing to give informed consent and agree to terms of the study
* Have assistance home; no driving for 24 hours

Exclusion Criteria:

* - Gestational ages 11 0/7 weeks or more
* Gestational age less than 6 0/7 weeks
* Incomplete abortion
* Premedication with misoprostol
* Use of narcotic pain or anti-anxiety medication within past 24 hours
* Use of heroin or methadone within last 3 months
* Chronic alcoholism or alcohol intoxication within past 24 hours
* Requested narcotics or Intravenous sedation (prior to randomization)
* Allergic reaction or allergy to cherry/cherry flavoring or lidocaine or non-steroidal anti-inflammatory drugs (NSAIDs)
* Allergic reaction or sensitivity to benzodiazepines including hyperactive or aggressive behavior (paradoxical reaction)
* Medical problem necessitating inpatient procedure
* Untreated acute cervicitis or pelvic inflammatory disease
* Known acute narrow-angle glaucoma
* Weighing less than 100 lb (45 kg)
* Use of potent medications interfering with microsomal metabolism within past 48 hours (carbamazepine (Tegretol), cimetidine (Tagamet), diltiazem (Cardizem), erythromycin, fluconazole (Diflucan), itraconazole (Sporanox), ketoconazole (Nizoral), phenobarbital, phenytoin (Dilantin), nelfinavir, ranitidine (Zantac), rifampin (Rifadin), ritonavir (Norvir), saquinavir, verapamil (Calan))

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bayer, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Planned Parenthood Columbia Willamette, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bayer LL, Edelman AB, Fu R, Lambert WE, Nichols MD, Bednarek PH, Miller K, Jensen JT. An Evaluation of Oral Midazolam for Anxiety and Pain in First-Trimester Surgical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):37-46. doi: 10.1097/AOG.0000000000000913. PMID 26241254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, placebo-controlled trial was conducted at Planned Parenthood Columbia/ Willamette in Portland, Oregon, between May 2013 and December 2013.
Period: Overall Study
Arm/Group | Midazolam and Ibuprofen | Placebo-cherry Syrup and Ibuprofen
Started | 62 | 62
Completed | 62 | 61
Not Completed | 0 | 1
Not completed — Changed decision to have an abortion | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject in the placebo group did not complete the study after changing mind to have abortion. Baseline information and characteristics on that subject was still collected and included where applicable in study outcomes and data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (5.3) | 25.5 (5.8) | 25.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 53 | 54 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 44 | 42 | 86
  More than one race | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Parity [Number; unit: participants]
  Nulliparous | 38 | 32 | 70
  Parous | 24 | 30 | 54
Previous vaginal deliveries [Number; unit: participants]
  Yes | 20 | 22 | 42
  No | 42 | 40 | 82
Previous surgical abortion [Number; unit: participants]
  Yes | 21 | 23 | 44
  No | 41 | 39 | 80
Level of menstrual symptoms [Number; unit: participants]
  Easy or mild cramping | 30 | 40 | 70
  Requiring medication or unable to attend work | 32 | 22 | 54
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.9 (6.0) | 25.9 (5.5) | 25.9 (5.7)
Self-reported depression [Number; unit: participants]
  Yes | 19 | 14 | 33
  No | 43 | 48 | 91
Self-reported anxiety [Number; unit: participants]
  Yes | 14 | 14 | 28
  No | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Subject Perception of Pain and Anxiety During Uterine Aspiration
Description: Subjects will be asked to rate anxiety and pain at the time of uterine aspiration by marking along a 100 mm Visual Analog Scale, with 0mm being No Pain/Anxiety and 100mm being Worst Imaginable Pain/Anxiety
Time Frame: at time of uterine aspiration (30-60 minutes after premedication)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
mm
  Pain with Aspiration | 74.3 (20.6) | 70.1 (22.1)
  Anxiety with Aspiration | 68.2 (28.1) | 60.9 (27.3)

2. Secondary Outcome: Subject Anticipated Perception of Pain and Anxiety During Uterine Aspiration at Baseline
Description: Subjects will be asked to rate their anticipated anxiety and pain at the time of uterine aspiration by marking along a mm Visual Analog Scale, with 0mm being No Pain/Anxiety and 100mm being Worst Imaginable Pain/Anxiety
Time Frame: Baseline (upon entry into study)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 62 | 62
mm
  Expected Anxiety | 77.5 (20.6) | 74.2 (20.1)
  Expected Pain | 67.2 (19.7) | 69.2 (17.8)

3. Secondary Outcome: Subject Perception of Pain and Anxiety Upon Entering Procedure Room
Description: Subjects will be asked to rate anxiety and pain upon entering procedure room by marking along a mm Visual Analog Scale, with 0mm being No Pain/Anxiety and 100mm being Worst Imaginable Pain/Anxiety
Time Frame: upon entering procedure room (30-60 minutes after premedication)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
mm
  Anxiety at Room Entry | 51.4 (25.4) | 34.5 (22.9)
  Pain at Room Entry | 17.5 (21.1) | 10.1 (15.4)

4. Secondary Outcome: Subject Perception of Pain and Anxiety Post Procedure
Description: Subjects will be asked to rate anxiety and pain 30 minutes post-operatively by marking along a mm Visual Analog Scale, with 0mm being No Pain/Anxiety and 100mm being Worst Imaginable Pain/Anxiety
Time Frame: 30 minutes post operatively
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
mm
  Anxiety Post Procedure | 20.9 (22.6) | 14.4 (13.5)
  Pain Post Procedure | 34.7 (23.3) | 37.1 (24.6)

5. Secondary Outcome: Subject Perception of Anxiety With Patient Positioning Procedure
Description: Subjects will be asked to rate anxiety prior to starting pelvic exam by marking along a mm Visual Analog Scale, with 0mm being No Anxiety and 100mm being Worst Imaginable Anxiety
Time Frame: prior to starting pelvic exam (30-60 minutes after premedication)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
mm | 56.6 (26.4) | 45.4 (26.3)

6. Secondary Outcome: Subject Perception of Pain During Cervical Dilation
Description: Subjects will be asked to rate pain at the time of cervical dilation by marking along a mm Visual Analog Scale, with 0mm being No Pain and 100mm being Worst Imaginable Pain
Time Frame: with cervical dilation (30-60 minutes after premedication)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
mm | 73.0 (21.2) | 69.3 (19.9)

7. Secondary Outcome: State-Trait Anxiety Inventory for Anxiety at Baseline
Description: To measure the mean State-Trait Anxiety Inventory (STAI) Form Y-1 for anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." Each type of anxiety has its own 4-point scale of 20 different questions that are scored. The 4-point scale for S-anxiety is as follows: 1.) not at all, 2.) somewhat, 3.) moderately so, 4.) very much so. The 4-point scale for T-anxiety is as follows: 1.) almost never, 2.) sometimes, 3.) often, 4.) almost always. Scores range from 20 to 80, with higher scores indicate greater anxiety. State anxiety items and Trait anxiety items were each summed in assessment to provide two total scores for each participant, a State anxiety score and a Trait anxiety score. Mean and standard deviation of total scores for each group are reported.
Time Frame: Baseline (upon entry into study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 62 | 62
units on a scale
  State anxiety level | 50.8 (11.0) | 51.3 (9.7)
  Trait anxiety level | 40.1 (10.8) | 38.6 (9.7)

8. Secondary Outcome: Patient Satisfaction With Pain and Anxiety 30 Minutes Postoperatively
Description: To assess whether oral midazolam is associated with differences in overall patient satisfaction with pain and anxiety control and abortion experience at 30 min postoperatively as measured by a mm Visual Analog Scale with 0mm being Not At All Satisfied and 100mm being Very Satisfied
Time Frame: 30 minutes post-operatively
Measure: Mean (Standard Deviation); unit: mm on a 100 mm Visual Analog Scale
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 61
mm on a 100 mm Visual Analog Scale
  Satisfaction with anxiety control (100-mm VAS) | 56.1 (29.6) | 68.9 (24.7)
  Satisfaction with pain control (100-mm VAS) | 43.2 (30.7) | 50.0 (27.3)

9. Secondary Outcome: Subject Satisfaction With Pain and Anxiety 1-3 Days Post Procedure
Description: To assess whether oral midazolam is associated with differences in overall patient satisfaction with pain and anxiety control and abortion experience at 1-3 days postoperatively as measured by a mm VAS with 0mm being Not At All Satisfied and 100mm being Very Satisfied
Time Frame: 1-3 days post-operatively
Measure: Mean (Standard Deviation); unit: mm on a 100 mm Visual Analog Scale
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 61
mm on a 100 mm Visual Analog Scale
  Satisfaction with anxiety control (100-mm VAS) | 50.2 (31.7) | 64.7 (28.2)
  Satisfaction with pain control (100-mm VAS) | 36.6 (30.8) | 48.2 (30.1)

10. Secondary Outcome: Subject Extent of Amnesia Using Amnesia Score
Description: To assess the extent of amnesia 30 min postoperatively as measured by ability to recall procedure using 4-point scale (0 = unable to recall any proportion of the procedure, 1 = able to recall and describe some portions of the procedure, but overall has minimal recall of the procedure, 2 = able to recall and describe most of the procedure, but admits to inability to recall some portion of the procedure, 3 = able to recall and describe the entire procedure).
Time Frame: 30 minutes postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 61
Participants
  Partial to complete amnesia (score 0,1,2) | 16 | 31
  No Amnesia (score 3) | 45 | 30

11. Secondary Outcome: Subject Extent of Amnesia
Description: To assess the extent of amnesia 1-3 days postoperatively as measured by 100mm Visual Analog Scale with 0mm being Remember Nothing and 100mm being Remember Everything.
Time Frame: 1-3 days postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 41 | 44
mm | 91.5 (12.8) | 61.3 (25.8)

12. Secondary Outcome: Subject Extent of Sedation
Description: Subject extent of sedation 30-60 minutes after premedication, just prior to procedure as measured by the 6-point Ramsay Scale (1 = patient anxious agitated, or restless; 2 = patient cooperative, oriented, and tranquil; 3 = patient asleep, responds to commands only; 4 = patient asleep, responds to gentle shaking, light glabellar tap, or loud auditory stimulus; 5 = patient asleep, responds to noxious stimuli such as firm nail bed pressure; 6 = patient asleep, has no response to firm nail bed pressure or other noxious stimuli)
Time Frame: 30-60 minutes after premedication
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
Participants
  1 | 11 | 10
  2 | 50 | 51
  3 | 0 | 1
  4 or greater | 0 | 0

13. Secondary Outcome: Subject Vital Signs (Heart Rate)
Description: Subject heart rate will be assessed for the duration of the procedure
Time Frame: intraoperatively (30-60 minutes after premedication)
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: bmp
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
bmp | 80 [51 to 126] | 78.5 [50 to 137]

14. Secondary Outcome: Subject Vital Signs (Heart Rate) 30 Minutes Postprocedure
Description: Subject vital signs (heart rate) will be assessed 30 minutes postoperatively
Time Frame: 30 minutes postoperatively
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
bpm | 70.1 (12.4) | 72 (11.8)

15. Secondary Outcome: Subject Nausea 30 Minutes Postprocedure
Description: Subject nausea will be assessed 30 minutes postoperatively using a 100mm Visual Analog Scale with 0mm being None and 100mm being Worst Imaginable
Time Frame: 30 minutes postoperatively
Measure: Mean (Full Range); unit: 100-mm visual analog sclae for nausea
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 61
100-mm visual analog sclae for nausea | 9.5 [0 to 80] | 3.5 [0 to 71]

16. Secondary Outcome: Subject's Correct Identification of Receiving Midazolam or Placebo
Description: Number of patient's who could correctly determine if they received study drug or placebo when asked
Time Frame: 30 minutes postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 61
Participants | 43 | 48

17. Secondary Outcome: Subject Vital Signs (Oxygenation Saturation)
Description: Subject oxygenation status will be assessed for the duration of the procedure
Time Frame: intraoperatively (30-60 minutes after premedication)
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
percent saturation | 98.3 (1.2) | 98.1 (1.0)

18. Secondary Outcome: Subject Vital Signs (Oxygenation Saturation) 30 Minutes Postprocedure
Description: Subject vital signs (oxygenation saturation) will be assessed 30 minutes postoperatively
Time Frame: 30 minutes postoperatively
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
percent saturation | 98.3 (1.2) | 98.1 (1.0)

19. Secondary Outcome: Subject Sleepiness 30 Minutes Postprocedure
Description: Subject sleepiness will be assessed 30 minutes postoperatively using a 100mm Visual Analog Scale with 0mm being None and 100mm being Worst Imaginable
Time Frame: 30 minutes postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Number analyzed (Participants) | 61 | 62
units on a scale | 40.1 (29.3) | 56.6 (24.6)

20. Secondary Outcome: Number of Participants With Need for Additional Postoperative Pain Medication
Description: Subjects will be assessed 30 minutes postoperatively for need of additional pain medications.
Time Frame: 30 minutes postoperatively
Population: One participant in the Midazolam group left the study. One participant in the placebo group decided not to have the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Ibuprofen | Placebo-cherry Syrup and Ibuprofen
Number analyzed (Participants) | 61 | 61
Participants
  Ondansetron | 3 | 2
  Hydrocodone/acetaminophen | 2 | 1

ADVERSE EVENTS:
Arm/Group | Placebo-cherry Syrup and Ibuprofen | Midazolam and Ibuprofen
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 2/62 | 3/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-cherry Syrup and Ibuprofen (N=62) | Midazolam and Ibuprofen (N=62)
Reaspiration (Surgical and medical procedures) | 2 (2) | 1 (1)
Cervical laceration (Surgical and medical procedures) | 0 (0) | 1 (1)
Hemorrhage (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No